CLINICAL TRIAL: NCT01504737
Title: Rehabilitation in the Form of Exercise Training in Aortic Stenosis Patients (RASP)
Brief Title: Rehabilitation in Aortic Stenosis Patients
Acronym: RASP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion rate, failure to recruit a priori determined no of patients.
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Kristofer Hedman, Principal Investigator, BSc, Physiotherapist, PhD-student, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RASP
Record Dates: First submitted 2012-01-02; First posted 2012-01-05 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Aortic Valve Stenosis
Keywords: Exercise; Physical Activity; Physiotherapy; Exercise test; Quality of Life; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Motor Activity | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised Exercise Training (Experimental): 12 weeks of 40 min aerobic bicycle ergometer exercise 3 times per week.
  Interventions: Other: Aerobic Exercise Training
- Physical Activity Recommendations (Active Comparator): Written and verbal information on minimal level of physical activity recommended.
  Interventions: Other: Physical Activity Recommendations

INTERVENTIONS:
Other: Aerobic Exercise Training — 12 weeks of endurance training, 40 minutes, 3 times per week on ergometer bicycle.
  Other Names: Physiotherapy; Physical activity
  Arms: Supervised Exercise Training
Other: Physical Activity Recommendations — Written and verbal information on minimal level of physical activity recommended.
  Other Names: Exercise
  Arms: Physical Activity Recommendations

SUMMARY:
SURVEY OF THE FIELD Aortic stenosis (AS) is the most common valve disease and increasing due to a growing elderly population. The therapy is aortic valve replacement (AVR). Studies on postoperative rehabilitation of AS pts are scarce. In the few studies available, a mix of valve diseases is presented without considering the differences in pathophysiology and the training regimes are not clearly described.

PURPOSE, AIMS & HYPOTHESIS The investigators purpose is to evaluate whether a supervised cardiac rehabilitation program improves the objective physical capacity and quality of life (QoL) of patients after AVR due to AS, and compare this to patients training by their own. The investigators hypothesize that supervised exercise training may be a more efficient way of rehabilitating these patients.

DESIGN This is a controlled randomized clinical trial comparing 12 weeks of supervised exercise training 3 times per week to home-based training based upon public health recommendations of minimum level of physical activity.

SIGNIFICANCE & IMPLEMENTATION Positive results would support that an organized program of exercise training improves physical capacity and QoL in AS patients following AVR with potential benefit for both patients and society.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery with aortic valve replacement for aortic stenosis at the thoracic surgery department at Linköping University hospital, Linköping.
* Geographical residence no further from hospital than permitting visit to Supervised Exercise Training 3 times per week

Exclusion Criteria:

* Any concommitant heart disease
* Other surgical intervention at time of valve replacement
* Age under 18 years
* Symptomatic lung disease
* Any disability or disease hampering participation in exercise training
* Cannot communicate with spoken Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake | Before (within one week before intervention), 1 week after and 12 months after intervention
  Physical capacity measured with cardiopulmonary exercise testing (CPET) on bicycle ergometer.

SECONDARY OUTCOMES:
Change in Health-related Quality of Life | Before (within one week before intervention), 1 week after and 12 months after intervention
  Short-form 36, version 2
Change in Physical activity level | Before (within one week before intervention), 1 week after and 12 months after intervention
  PAL - Physical activity level, measured with International Physical Activity Questionnary (IPAQ)
Change in hs-CRP | Before (within one week before intervention), 1 week after and 12 months after intervention
Change in NT-pro-BNP | Before (within one week before intervention), 1 week after and 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eva Nylander, PhD, Study Director — Linkoeping University
Locations (1):
- Heart and Medicine Center, Linköping University Hospital, Linköping, Östergötland County, Sweden